CLINICAL TRIAL: NCT03751020
Title: Development and Preliminary Trial of a Brief, Portable Health Intervention for Rural Sexual Minority Emerging Adults
Acronym: Project LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1512016952; 1R21MH113860-01 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-11-23 (Actual); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Depression; Suicidality; Substance Abuse; HIV; Minority Stress
Keywords: Expressive Writing; Minority Stress; Lesbian Gay Bisexual
MeSH Terms: conditions — Depression; Suicidal Ideation; Substance-Related Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expressive Writing (EW) (Experimental): Expressive Writing (EW) prompts individuals to write about personally stressful events, potentially enabling cognitive processing of unresolved, psychological and physiological stressors.
  Interventions: Behavioral: Expressive Writing (EW) Intervention
- Self-Affirmation (SA) (Experimental): Self-Affirmation (SA) interventions prompt individuals to write advice to a (hypothetical) similarly stigmatized person regarding how best to cope with stigma-related stress. By affirming one's own stigmatized identity through the process of helping another similarly stigmatized person.
  Interventions: Behavioral: Self-Affirmation (SA) Intervention
- Control (Placebo Comparator): Participants randomly assigned to the control condition will be asked to write about what they have done since waking up that morning for 20 minutes across 3 consecutive days.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Expressive Writing (EW) Intervention — The EW intervention will utilize the procedures piloted earlier with gay and bisexual male college students in urban and rural regions of the US. In this condition, participants will be instructed to write for 20 minutes across three consecutive days in a free-form manner about the most stressful or traumatic LGB-related event that they have encountered.
  Arms: Expressive Writing (EW)
Behavioral: Self-Affirmation (SA) Intervention — The SA intervention will ask participants to read a brief description, over the course of 3 consecutive days, of a (hypothetical) LGB youth who is facing minority stress. Each day's description will contain a different LGB youth facing a different stigma-related stressor derived from Phase 1 and 2 interviews. Participants will then be asked to write a letter for 20 minutes to advise the LGB youth how best to cope with minority stress drawing on their personal experiences.
  Arms: Self-Affirmation (SA)
Other: Control — Participants randomly assigned to the control condition will be asked to write about what they have done since waking up that morning for 20 minutes across 3 consecutive days. This control matches the time and activity of the EW and SA arms and has been implemented across dozens of EW and SA studies.
  Arms: Control

SUMMARY:
The purpose of this study is to test the feasibility of writing interventions specifically designed for lesbian, gay, and bisexual (LGB) emerging adults (ages 18-29) that are aimed at improving the outcomes: depression, suicidality, substance abuse and HIV risk behaviors.

DETAILED DESCRIPTION:
This study is considered the third part ("Phase 3") of a larger study where parts one and two were designed to utilize elicitation focus groups to develop effective intervention materials (Phase 1) and then refine the developed materials through structured interviews (Phase 2). Phase 3 will test feasibility and assess early signs of efficacy of writing interventions. To do this, participants will be randomized to one of three arms (one arm will serve as control). Those that choose to participate will be asked to complete outcome measures (depressive symptoms, suicidality, use of alcohol and illicit drugs, HIV risk behavior) and measures of proposed mediators (self-reported and biological stress, behavioral and emotional self-regulation) and moderators (e.g., social support, identity centrality) at baseline, post-intervention, and three-month follow-up. In addition, structured interviews with 15 intervention participants will be used to refine study procedures as the investigators scale up this intervention for a future randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as lesbian, gay, or bisexual
* Live in Washington county, Tennessee (TN), or any of its 6 contiguous counties in northeastern TN
* Have personal Internet access
* Hair at least 2cm in length

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - College of the Holy Cross, Worcester, Massachusetts
  - East Tennessee State University, Johnson City, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion for three years.
Access Criteria: Data access requests from qualified academic investigators for non-commercial research interests will be reviewed by study investigators. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Derived] Pachankis JE, Williams SL, Behari K, Job S, McConocha EM, Chaudoir SR. Brief online interventions for LGBTQ young adult mental and behavioral health: A randomized controlled trial in a high-stigma, low-resource context. J Consult Clin Psychol. 2020 May;88(5):429-444. doi: 10.1037/ccp0000497. PMID 32271053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were specifically recruited through tailored advertising on geo-targeted websites; bulletin boards and listservs of local colleges; in-person announcement and flyers at local businesses, community events, and the gay-straight alliances of area schools. Participants completed a brief online survey to confirm eligibility.
Pre-assignment Details: Participants completed a brief online survey to confirm eligibility, defined as:
  age 18 -29; identifying as sexual minority; currently living in one of the eligible counties; and having daily personal Internet access. Participants emailed a photo of an identification card(e.g. a driver's license), as proof of age. 108 people were randomized.
Period: Overall Study
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Started | 36 | 36 | 36
Post Intervention | 33 | 33 | 30
3 Month Follow Up | 27 | 32 | 26
Completed | 27 | 32 | 26
Not Completed | 9 | 4 | 10
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 7 | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA) | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.14 (3.24) | 23.47 (2.88) | 23.42 (3.25) | 23.68 (3.11)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity.
  Participants
    Man | 10 | 12 | 9 | 31
    Woman | 20 | 21 | 19 | 60
    Transgender Man | 1 | 3 | 3 | 7
    Transgender Woman | 1 | 0 | 0 | 1
    Gender Queer | 4 | 2 | 4 | 10
    Gender Non-Conforming/Binary | 3 | 3 | 4 | 10
    Two-spirit | 0 | 0 | 1 | 1
    Other | 2 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth.
  Participants
    Female | 25 | 26 | 26 | 77
    Male | 11 | 10 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 35 | 36 | 35 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race (choose all that apply)
  Participants
    American Indian /Alaskan Native | 0 | 2 | 0 | 2
    Asian | 1 | 0 | 0 | 1
    Black/African American | 2 | 4 | 4 | 10
    Native Hawaiian/Pacific Islander | 1 | 0 | 0 | 1
    White | 33 | 33 | 34 | 100
    Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 36 | 108
Sexual Orientation [Count of Participants; unit: Participants]
  Asexual | 0 | 1 | 1 | 2
  Bisexual | 13 | 9 | 8 | 30
  Gay | 8 | 9 | 9 | 26
  Lesbian | 12 | 9 | 9 | 30
  Pansexual | 3 | 6 | 6 | 15
  Questioning | 0 | 0 | 1 | 1
  Other | 0 | 2 | 2 | 4
Education Level [Count of Participants; unit: Participants]
  Less than College | 18 | 19 | 21 | 58
  College Degree | 18 | 17 | 15 | 50
Employment Status [Count of Participants; unit: Participants]
  Full-time | 14 | 13 | 14 | 41
  Part-time | 21 | 13 | 12 | 46
  Student | 0 | 5 | 6 | 11
  Unemployed | 1 | 5 | 4 | 10
Personal Income [Count of Participants; unit: Participants] — Income for the last calendar year.
  Participants
    Less than $10,000 | 11 | 17 | 13 | 41
    More than $10,000 | 25 | 19 | 23 | 67
Family Class Background [Count of Participants; unit: Participants] — Description of social class/socioeconomic background.
  Participants
    Poor | 3 | 7 | 6 | 16
    Working Class | 12 | 11 | 13 | 36
    Lower Middle Class | 8 | 4 | 5 | 17
    Middle Class | 10 | 11 | 11 | 32
    Upper Middle Class | 3 | 3 | 1 | 7
Relationship Status [Count of Participants; unit: Participants]
  Single | 11 | 10 | 14 | 35
  In a Relationship | 25 | 26 | 22 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression.
Description: Depression will be measured using the Center for Epidemiological Studies -- Depression Scale (CESD). An overall depression score is computed as the sum of 20 items, with items 3, 11, 14, and 16 reversed. In cases with internally missing data (items not answered), the sums are computed after imputation of the missing values: # items on scale / # actually answered, multiplied by the sum obtained from the answered items. A range of 0-60, with higher scores indicating more depressive symptomatology during the past week.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 24.75 (11.83) | 25.17 (12.07) | 29.06 (13.41)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 21.03 (11.79) | 17.42 (11.46) | 21.73 (13.45)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 23.44 (13.09) | 18.45 (10.97) | 22.92 (14.61)
Statistical Analysis 1: Comparison: Control vs Expressive Writing (EW); The primary comparison was between EW and control to test the interaction between treatment and time; Test type: Superiority; p < 0.01, Mixed Models Analysis; Mean Difference (Net) = -6.34, 95% CI 2-sided [-11.03 to -1.64]

2. Primary Outcome: Change in Psychological Distress.
Description: Psychological Distress will be measured using the Brief Symptom Inventory (BSI). The BSI consists of 18 items scored 0-4. Items are averaged to yield a final score of 0-4. The higher the score, the greater the psychological distress.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 2.31 (0.85) | 2.22 (0.73) | 2.63 (0.86)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 1.84 (0.77) | 1.82 (0.67) | 2.08 (0.86)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 2.14 (0.92) | 1.77 (0.65) | 2.35 (0.80)
Statistical Analysis 1: Comparison: Control vs Expressive Writing (EW); The primary comparison was between EW and control to test the interaction between treatment and time; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.62 to -0.03]

3. Primary Outcome: Change in Anxiety.
Description: Anxiety will be measured using the Beck Anxiety Inventory (BAI). The BAI total score is reported, which is the sum of all 21 items; with no subscales. The range of scores is 0-63, with higher scores indicating higher anxiety.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 21.72 (14.14) | 20.28 (12.29) | 26.94 (13.91)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 14.73 (13.43) | 13.54 (10.91) | 19.47 (13.16)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 18.26 (13.19) | 13.03 (10.55) | 19.73 (10.78)
Statistical Analysis 1: Comparison: Control vs Expressive Writing (EW); The primary comparison was between EW and control to test the interaction between treatment and time; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -4.03, 95% CI 2-sided [-8.55 to 0.47]

4. Primary Outcome: Change in Suicidality - Suicidal Ideation.
Description: Suicidal ideation will be measured using the Suicidal Ideation Attributes Scale (SIDAS) . Total SIDAS scores are calculated as the sum of the five items, with controllability reverse scored (10=0, 9=1, …, 0=10). Total scores range from 0 to 50.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 6.05 (9.81) | 4.19 (6.92) | 9.42 (11.21)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 2.36 (4.08) | 1.21 (3.57) | 2.70 (6.24)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 4.63 (8.19) | 3.87 (7.40) | 5.31 (7.54)
Statistical Analysis 1: Comparison: Control vs Expressive Writing (EW); The primary comparison was between EW and control to test the interaction between treatment and time; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Net) = 1.12, 95% CI 2-sided [-6.48 to 8.77]

5. Primary Outcome: Change in Alcohol Use.
Description: Alcohol use in participants will be assessed using the Alcohol Use Disorders Identification (AUDIT) instrument. The AUDIT consists of 10 items. Each of the questions has a set of responses to choose from, and each response has a score ranging from 0 to 4. All response scores should be added and recorded as "Total". Total scores of 8 or more are recommended as indicators of hazardous and harmful alcohol use, as well as possible alcohol dependence. (A cut-off score of 10 will provide greater specificity but at the expense of sensitivity.) The score range is 0-40. Higher scores indicate greater hazardous drinking.
Time Frame: Baseline, Post Intervention, 3 Months
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 5.08 (3.77) | 4.25 (4.29) | 5.97 (6.00)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 4.67 (4.00) | 3.70 (4.33) | 3.73 (4.35)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 5.26 (4.62) | 2.91 (3.76) | 5.58 (5.98)
Statistical Analysis 1: Comparison: Control vs Expressive Writing (EW); The primary comparison was between EW and control to test the interaction between treatment and time; Test type: Superiority; p = 0.10, Mixed Models Analysis; Mean Difference (Net) = -1.28, 95% CI 2-sided [-2.80 to 0.24]

6. Primary Outcome: Change in Drug Use.
Description: The Short Inventory of Problems-Modified for Drug Use (SIP-DU) is a 15-item scale that asks respondents to rate each item on a dichotomous scale ("No" = 0, "Yes" = 1). Total score reported, which is the sum of all items; no subscales: Range 0-15, higher scores indicate greater problems with drug use.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 0.39 (0.99) | 0.31 (0.98) | 1.47 (2.99)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 0.36 (1.03) | 0.67 (2.53) | 0.57 (1.70)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 0.33 (0.83) | 0.84 (2.89) | 1.58 (3.56)
Statistical Analysis 1: Comparison: Control vs Expressive Writing (EW); The primary comparison was between EW and control to test the interaction between treatment and time; Test type: Superiority; p = 0.76, Mixed Models Analysis; Mean Difference (Net) = 0.09, 95% CI 2-sided [-1.19 to 1.57]

7. Primary Outcome: Suicidal Intent
Description: Suicidal intent will be assessed using a single item that asks: Within the last 3 months/past week, have you seriously considered attempting suicide? [yes/no] Number of participants who reported suicidal intent is reported. Originally titled "Change in Suicidality - Suicidal Thoughts".
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Baseline | 4 | 4 | 9
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 0 | 0 | 1
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 3 | 1 | 2

8. Primary Outcome: Attempted Suicide
Description: Suicide attempts will be assessed using a single item that asks: Within the last past 3 months/past week, have you actually attempted suicide? [yes/no]. Reported are the number of participants who reported that they had attempted suicide. Original title: "Change in Suicidality: Suicide Attempts".
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Baseline | 1 | 0 | 1
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 0 | 0 | 0
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 0 | 0 | 0

9. Secondary Outcome: Self Injury.
Description: Self injury behaviors will be assessed with the item that asks: How many times in the past 3 months/past week have you engaged in self-harm behavior (e.g., cutting, biting, burning, hitting self) with the intent of harming, but not killing, yourself? Reported are the frequency of self-harm behaviors/self-injury reported by participants. Original title: "Change in Self Injury".
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: self-harm behaviors
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
self-harm behaviors
  Baseline | 0.61 (1.50) | 1.36 (5.11) | 0.94 (2.11)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 0.12 (0.48) | 0.21 (1.22) | 0.07 (0.25)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 0.26 (0.71) | 0.97 (4.45) | 1.27 (3.97)

10. Secondary Outcome: Rumination
Description: Rumination will be assessed using the Ruminative Response Scale - Brooding Subscale (RRS). This scale is modified from the original measure where only items 5, 10, 13, 15 and 16 are used. Each item is scored by respondents on a scale of 1 to 4. To get the overall score, the 5 items are summed; total scores range from 5-20, with higher scores indicating greater brooding and rumination (related to depression) in an individual.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 12.39 (3.68) | 12.97 (3.48) | 13.03 (3.55)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 11.58 (3.57) | 11.67 (3.48) | 12.10 (4.41)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 11.44 (4.86) | 10.81 (3.81) | 11.81 (3.62)

11. Secondary Outcome: Perceived Support
Description: Perceived social support is measured using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12 item instrument that uses a scale 1-7 to rate each item. The scoring is done by taking the average of the items- therefore a score of 7 indicates the highest level of perceived social support.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 5.11 (1.30) | 5.35 (0.94) | 4.89 (1.40)
  Post-Intervention: number analyzed (Participants) | 36 | 33 | 30
  Post-Intervention | 5.10 (1.08) | 5.34 (0.93) | 5.03 (1.44)
  3 Months: number analyzed (Participants) | 36 | 32 | 26
  3 Months | 5.12 (1.39) | 5.53 (1.01) | 5.09 (1.65)

12. Secondary Outcome: Hopelessness
Description: Hopelessness will be measured using the Beck Hopelessness Scale (BHS). The BHS is a 20-item dichotomous scale ("No" = 0, "Yes" = 1). Items 1, 3, 5, 6, 8, 10, 13, 15 and 19 are reverse-scored. The total score is out of 20, where 20 would be the highest score and considered a negative indicator of hopelessness.
Time Frame: Baseline, Post Intervention, 3 Months
Population: Data analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 7.00 (6.08) | 5.14 (4.28) | 7.44 (6.07)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 6.93 (6.31) | 4.88 (4.87) | 7.80 (6.51)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 5.85 (5.80) | 5.19 (5.07) | 7.77 (7.00)

13. Secondary Outcome: Lesbian, Gay, Bisexual (LGB) Identity
Description: LGB identity will be measured using the 'LGB Identity Centrality' instrument.The measure consists of 4 items that are rated on a scale of 1-7. The summed scores have a range of 4-28 and the higher score would indicate a stong agreement (positive) with the centrality of one's LGB identity.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 22.44 (6.08) | 18.47 (5.36) | 20.11 (5.67)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 19.91 (5.17) | 17.33 (5.95) | 18.27 (7.08)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 20.74 (4.92) | 17.00 (5.81) | 18.27 (7.48)

14. Secondary Outcome: Change in Cortisol
Description: Participants will provide 50-100 hair strands (at least 2 cm in length) to be used to determine levels of stress based on the cortisol levels found in the analyses of the hair provided.
Time Frame: 1 and 4 months post baseline.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: pg/mg
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
pg/mg
  1 Month | 10.12 (12.20) | 8.28 (10.96) | 10.91 (15.85)
  4 Months: number analyzed (Participants) | 27 | 32 | 26
  4 Months | 10.37 (10.18) | 6.18 (5.49) | 12.21 (28.72)

15. Secondary Outcome: Change in Stress
Description: Stress will be assessed using the Perceived Stress Scale (PSS). Participants were asked to respond to the 14-item version. Participants respond to each item on a 0-4 scale and scores are obtained by reversing responses to the 7 positively stated items (items 4,5,6,7,9,10, & 13), and then summing across all scale items. Range = 0-56. Higher scores indicating higher perceived stress.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 30.25 (8.62) | 29.53 (8.40) | 31.61 (9.51)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 27.03 (9.96) | 24.70 (9.67) | 26.73 (8.58)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 28.41 (10.66) | 25.88 (7.77) | 28.69 (9.01)

16. Secondary Outcome: Change in Impulsiveness Total Score
Description: Impulsiveness will be assessed using the Barratt Impulsiveness Scale (BIS). The BIS is a 30 item questionnaire that uses a 1-4 rating scale per item. The 30-item self-report questionnaire, can yield a total score where the range is 30-120. The highest score indicates the greatest the level of impulsiveness.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 53.75 (11.92) | 51.03 (11.31) | 54.31 (4.11)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 52.35 (10.50) | 52.76 (12.34) | 54.06 (11.36)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 53.39 (11.38) | 54.14 (11.43) | 53.58 (9.37)

17. Secondary Outcome: Change in Impulsiveness- Attentional
Description: Impulsiveness will be assessed using the Barratt Impulsiveness Scale (BIS). The BIS is a 30 item questionnaire that uses a 1-4 rating scale per item. The 30-item self-report questionnaire, can yield a total score, as well as three factors: attentional (6, 5, 9, 11, 20, 24, 26, 28; motor (2, 3, 4, 16, 17, 19, 21, 22, 23, 25, 30); non-planning (1, 7, 8, 10, 12, 13, 14, 15, 18, 27, 29). The attentional scale has a range of 8-32, the greater the value, the greater the level of attentional impulsiveness.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 16.36 (4.98) | 16.44 (4.59) | 16.33 (4.11)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 15.79 (4.69) | 15.64 (4.62) | 16.70 (4.19)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 15.43 (4.33) | 15.75 (4.19) | 16.69 (5.53)

18. Secondary Outcome: Change in Impulsiveness- Motor
Description: Impulsiveness will be assessed using the Barratt Impulsiveness Scale (BIS-11). The BIS-11 is a 30 item questionnaire that uses a 1-4 rating scale per item. The 30-item self-report questionnaire, can yield a total score, as well as three factors: attentional (6, 5, 9, 11, 20, 24, 26, 28; motor (2, 3, 4, 16, 17, 19, 21, 22, 23, 25, 30); non-planning (1, 7, 8, 10, 12, 13, 14, 15, 18, 27, 29). The motor scale has a range of 11-44, the greater the value, the greater the level of motor impulsiveness.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 20.78 (4.33) | 20.78 (4.00) | 21.39 (4.14)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 15.71 (5.01) | 20.52 (3.94) | 21.23 (4.16)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 21.96 (5.17) | 21.23 (4.18) | 20.27 (3.11)

19. Secondary Outcome: Change in Impulsiveness- Non-Planning
Description: Impulsiveness will be assessed using the Barratt Impulsiveness Scale (BIS-11). The BIS-11 is a 30 item questionnaire that uses a 1-4 rating scale per item. The 30-item self-report questionnaire, can yield a total score, as well as three factors: attentional (6, 5, 9, 11, 20, 24, 26, 28; motor (2, 3, 4, 16, 17, 19, 21, 22, 23, 25, 30); non-planning (1, 7, 8, 10, 12, 13, 14, 15, 18, 27, 29). The non-planning scale has a range of 11-44, the greater the value, the greater the level of non-planning impulsiveness.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 17.00 (5.20) | 16.80 (5.59) | 16.58 (5.18)
  Post-Intervention: number analyzed (Participants) | 30 | 33 | 30
  Post-Intervention | 15.71 (5.01) | 16.61 (6.58) | 16.13 (5.31)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 16.00 (4.74) | 17.16 (6.06) | 16.62 (4.98)

20. Secondary Outcome: Change in Risk Taking
Description: Risk taking impulse will be assessed using the Columbia Card Task. Participants are presented with 32 face-down cards. Some of these cards are "gain cards" (which add either +10 or +30 points to the participant's total score) and some of these cards are "loss cards" (which subtract either -250 or -750 points from the participant's total score). On each trial, the participant may turn over as many cards as desired until a loss card is encountered or the participant chooses to not turn over any more cards. As a participant turns over more cards, the probability of encountering a loss card increases. Therefore, turning over more cards constitutes greater risk taking.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: This outcome measure was never collected.
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Change in Minority Stress (Rejection)
Description: To assess rejection as a form of minority stress, the Gay-Related Rejection Sensitivity Scale (GRRS) will be used.The Gay-related rejection sensitivity scale was adapted for this study to be gender-inclusive and has 12 items. Scale range 1-36, where higher scores indicate greater rejection sensitivity based on one's sexual orientation (worse outcome).
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 14.47 (7.35) | 12.33 (6.11) | 14.94 (7.43)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 12.92 (8.23) | 10.95 (6.51) | 12.99 (6.41)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 12.17 (8.16) | 9.31 (7.60) | 12.33 (5.65)

22. Secondary Outcome: Change in Parental Attitudes
Description: The participant's perception of their parent's attitudes towards their sexual orientation are assessed using the Parental Attitudes Toward Child's Sexual Orientation. This tool has 4 items- 2 that deal with mother/parent 1/closest female guardian, 2 that deal with father/parent 2/closest male guardian. The second item for each parent asks about their attitude towards the respondent's sexual orientation on a scale from 1 (completely tolerant and accepting) to 7 (completely hostile and rejecting). Scores for maternal and paternal attitude should be averaged for each participant. The score has a range from 1-7, where higher scores indicate greater rejection from parents (worse outcome).
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzes as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 2.85 (1.50) | 2.59 (1.52) | 2.61 (1.46)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 2.71 (1.21) | 2.60 (1.47) | 2.36 (1.28)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 2.75 (1.46) | 2.63 (1.36) | 2.68 (1.48)

23. Secondary Outcome: Change in Outness
Description: Participants openness about one's sexual orientation will be assessed using the Outness Inventory (OI). A respondent is asked to rate how open they are with various people in society (from family to strangers) on an 11 item questionnaire. The scale for responding is 0-7- where 7 indicates that a person is completely open with their sexual orientation status. The scale score is obtained by averaging the 11 items for a score range of 0-7, where higher scores indicate more openness about respondents' sexual orientation in different domains of their lives/different people. 0 indicates that an item does not apply/ there is no such group of people/person in the respondents' life. A score of 7 would indicate that one is completely open or "out" with respect to sexual orientation.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 4.46 (1.56) | 5.32 (1.43) | 5.05 (1.40)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 4.55 (1.66) | 5.13 (1.39) | 4.94 (1.21)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 4.95 (1.49) | 5.16 (1.49) | 5.01 (1.33)

24. Secondary Outcome: Change in Internalized Homophobia
Description: Internalized homophobia in participants will be assessed using the Internalized Homophobia Scale (IHS). The IHS score is obtained by averaging the scores across the 9 items (rather than summing). Range is 1-4, with higher scores indicating higher internalized stigma related to one's sexual orientation.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 1.42 (0.57) | 1.38 (0.50) | 1.58 (0.65)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 1.27 (0.64) | 1.27 (0.53) | 1.56 (0.58)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 1.29 (0.63) | 1.39 (0.57) | 1.52 (0.58)

25. Secondary Outcome: Change in Discrimination - 9 Items (Part 1)
Description: Everyday discrimination experienced by participants will be measured using the Everyday Discrimination - Sexual Orientation (EDSO) Part 1. Part 1 is a 9 item inventory where respondents rate statements on a scale of 1-6. The scale has a summed total score ranging from 9-54, higher scores indicate higher discrimination. The higher the score, the greater the feeling that one is discriminated against for one's sexual orientation.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 19.75 (10.63) | 19.22 (7.26) | 21.14 (8.72)
  Post Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post Intervention | 18.61 (9.47) | 17.88 (7.27) | 20.47 (9.42)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 17.81 (9.22) | 16.87 (7.49) | 17.81 (8.64)

26. Secondary Outcome: Change in Discrimination - Item 1 (Part 2)
Description: Everyday discrimination experienced by participants will be measured using the Everyday Discrimination - Sexual Orientation (EDSO) Part 2. Part 2 is a 2 item inventory where respondents rate statements on a scale of 0-3. The lower the score, the less the feeling that one is discriminated against overall for one's sexual orientation.
  Item 1: Overall, how much has discrimination based on your sexual orientation interfered with you having a full and productive life?
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 0.78 (0.76) | 0.89 (0.82) | 1.19 (0.98)
  Post Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post Intervention | 0.67 (0.66) | 1.00 (0.79) | 0.97 (0.89)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 0.74 (0.81) | 0.87 (0.72) | 0.73 (0.87)

27. Secondary Outcome: Change in Discrimination - Item 2 (Part 2)
Description: Everyday discrimination experienced by participants will be measured using the Everyday Discrimination - Sexual Orientation (EDSO) Part 2. Part 2 is a 2 item inventory where respondents rate statements on a scale of 0-3. The lower the score, the less the feeling that one is discriminated against overall for one's sexual orientation.
  Item 2: Overall, how much harder has your life been because of discrimination based on your sexual orientation?
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 1.03 (0.81) | 1.42 (0.87) | 1.53 (0.91)
  Post Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post Intervention | 1.00 (0.79) | 1.24 (0.87) | 1.30 (1.02)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 0.85 (0.72) | 1.06 (0.73) | 1.15 (0.97)

28. Secondary Outcome: Change in Victimization
Description: Feelings of victimization are captured using the LGBT Victimization Experiences measure. This questionnaire consists of 10 items. The LGBT victimization scale is rated on a 0 "Never" to 3 "3+ times" scale with a total score range 0-30. The total score reflects the amount of victimization one has experienced due to being known or thought to be LGBTQ. Higher scores indicate more negative experiences.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 1.47 (2.16) | 1.33 (2.05) | 2.56 (5.42)
  Post-Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post-Intervention | 0.30 (0.81) | 0.24 (0.56) | 0.67 (1.65)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 0.81 (1.33) | 0.97 (2.47) | 1.08 (2.42)

29. Secondary Outcome: Change in Religious Affiliation
Description: Tolerance of one's sexual orientation through the lense of one's practiced religion is measured using a single question. Respondents use a 1-7 scale to rate the question "How tolerant is your religion toward your sexual orientation?"- where 7 indicates total rejection and hostility.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 2.70 (1.86) | 3.05 (1.84) | 2.78 (2.06)
  Post Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post Intervention | 2.78 (1.57) | 2.79 (1.65) | 2.71 (1.94)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 2.20 (1.47) | 2.56 (1.50) | 3.13 (1.96)

30. Secondary Outcome: Change in Religious Strain
Description: Religious Strain Scale total score obtained by reverse scoring items 1-7 and then summing across the 20 items (range 0-60), higher scores indicate greater religious strain.
Time Frame: Baseline, Post Intervention (day 5), and 3 Months.
Population: Data were analyzed as intention to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Baseline | 29.08 (8.92) | 27.11 (10.01) | 32.75 (9.36)
  Post Intervention: number analyzed (Participants) | 33 | 33 | 30
  Post Intervention | 27.52 (9.52) | 26.52 (9.49) | 31.40 (10.62)
  3 Months: number analyzed (Participants) | 27 | 32 | 26
  3 Months | 27.11 (9.63) | 25.44 (9.31) | 29.50 (9.61)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for up to 3 months.
Arm/Group | Control | Expressive Writing (EW) | Self-Affirmation (SA)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT03751020/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT03751020/SAP_001.pdf